CLINICAL TRIAL: NCT06370806
Title: Interdisciplinary Weight Loss and Lifestyle Intervention for Obstructive Sleep Apnea in Women: The INTERAPNEA-Women Clinical Trial
Brief Title: Lifestyle Intervention for Obstructive Sleep Apnea in Women
Acronym: INTERAPNEA-W
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Fundación BBVA (Unknown); Universidad Loyola Andalucia (Other)
Responsible Party: Principal Investigator, Almudena Carneiro Barrera, Principal Investigator, Universidad Loyola Andalucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERAPNEA-Women
Record Dates: First submitted 2024-03-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants from the usual care group will not receive any type of intervention apart from the usual care (CPAP).
- Lifestyle Intervention (Experimental): Participants from this group will receive a interdisciplinary intervention addressing weight loss and lifestyle change including nutritional behavior change, aerobic exercise, sleep hygiene, and alcohol and tobacco cessation combined with usual care (i.e., CPAP)
  Interventions: Behavioral: Weight loss and lifestyle intervention

INTERVENTIONS:
Behavioral: Weight loss and lifestyle intervention — Interdisciplinary intervention addressing weight loss and lifestyle change including nutritional behavior change, aerobic exercise, sleep hygiene, and alcohol and tobacco cessation combined with usual care (i.e., CPAP)
  Arms: Lifestyle Intervention

SUMMARY:
Obesity is a major risk factor for obstructive sleep apnoea (OSA), the most common sleep-disordered breathing related to neurocognitive and metabolic syndromes, type II diabetes, and cardiovascular diseases. Although strongly recommended for this condition, there are no studies on the effectiveness of an interdisciplinary weight loss and lifestyle intervention including nutrition, exercise, sleep hygiene, and smoking and alcohol cessation in women. INTERAPNEA-Women is a randomized controlled trial with a two-arm parallel design aimed at determining the effects of an interdisciplinary tailored weight loss and lifestyle intervention on OSA outcomes. The study will include 180 females aged 18-65 with a body mass index of ≥25 kg/m2 and severe to moderate OSA randomly assigned to usual care (i.e., continuous positive airway pressure), or interdisciplinary weight loss and lifestyle intervention combined with usual care. Outcomes will be measured at baseline, intervention end-point, and six-month post-intervention, including apnoea-hypopnoea index (primary outcome), other neurophysical and cardiorespiratory polysomnographic outcomes, sleep quality, daily functioning and mood, body weight and composition, physical fitness, blood biomarkers, and health-related quality of life. INTERAPNEA may serve to establish a cost-effective treatment not only for the improvement of OSA and its vast and severe comorbidities, but also for a potential remission of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Previous clinical diagnosis of moderate/severe OSA (AHI > 15)
* Female patients aged between 18-65 years.
* Body mass index > 25 kg/m2.
* Use of CPAP.
* Motivation to participate in the study.
* Signed informed consent form.

Exclusion Criteria:

* Sleep disorder other than OSA.
* Clinically significant psychiatric, neurological, or medical disorders other than OSA.
* Use of prescription drugs or clinically significant drugs affecting sleep.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Apnoea-hypopnoea index (AHI) | Post-intervention (2 months)
  Change in apnea (airflow reduction greater than or equal to 90%) and hypopnea (airflow reduction greater than or equal to 30%) episodes per hour of sleep measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)

SECONDARY OUTCOMES:
Oxygen desaturation index (ODI) | Post-intervention (2 months)
  Change in the number of oxygen desaturations greater than or equal to 4%/h measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Oxygen saturation (SaO2) mean | Post-intervention (2 months)
  Change in the average of oxygen saturation measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Oxygen saturation (SaO2) nadir | Post-intervention (2 months)
  Minimum oxygen saturation measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Sleep efficiency | Post-intervention (2 months)
  Change in the total sleep time/total time in bed measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Light sleep (N1 and N2 stages) | Post-intervention (2 months)
  Change in the percentage of light sleep (N1 and N2 stages) measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Deep sleep (N3 stage) | Post-intervention (2 months)
  Change in the percentage of deep sleep (N3 stage) measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Rapid eye movement (REM) sleep | Post-intervention (2 months)
  Change in the percentage of REM sleep measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Excessive daytime sleepiness (EDS) | Post-intervention (2 months)
  Change in the difficulty in maintaining a desired level of wakefulness, measured by the Epworth sleepiness scale (ESS) from baseline to post-intervention. ESS is a 4-point scale (0 = no chance of dozing, 1 = slight chance of dozing, 2 = moderate chance of dozing, 3 = high chance of dozing) that measures the usual chances of dozing off or falling asleep while engaged in eight different activities. An ESS total score from 0 to 9 is considered to be normal while an ESS total score > 9 indicates high daytime sleepiness.
Sleep Quality | Post-intervention (2 months)
  Change in Pittsburgh Sleep Quality Index (PSQI) from baseline to post-intervention. This scale includes a total of 19 self-rated items combined to form seven component scores i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction), each of which has a range of 0-3 points. The sum of these seven PSQI component scores is considered to obtain a global PSQI score (ranging from 0-21), with higher scores indicating poorer sleep quality.
Wake After Sleep Onset (WASO) | Post-intervention (2 months)
  Change in Wake After Sleep Onset (WASO; minutes) measured by a respiratory polygraphy, from baseline (week 0) to post-intervention (2 months)
Fat mass (kg) | Post-intervention (2 months)
  Change in fat mass (kg) measured by a whole-body densitometry using dual-energy X-ray absorptiometry (DEXA), from baseline (week 0) to post-intervention (2 months)
Visceral adipose tisue (g) | Post-intervention (2 months)
  Change in visceral adipose tisue (g) measured by a whole-body densitometry using dual-energy X-ray absorptiometry (DEXA), from baseline (week 0) to post-intervention (2 months)
Body weight (kg) | Post-intervention (2 months)
  Change in body weight (kg) measured by a scale from baseline (week 0) to post-intervention (2 months)
Neck circumference (cm) | Post-intervention (2 months)
  Change in neck circumference (cm) measured by a tape measure from baseline (week 0) to post-intervention (2 months)
Chest circumference (cm) | Post-intervention (2 months)
  Change in chest circumference (cm) measured by a tape measure from baseline (week 0) to post-intervention (2 months)
Waist circumference (cm) | Post-intervention (2 months)
  Change in waist circumference (cm) measured by a tape measure from baseline (week 0) to post-intervention (2 months)
Mean blood pressure (mm HG) | Post-intervention (2 months)
  Change in mean blood pressure (mm HG) measured by a blood pressure cuff from baseline (week 0) to post-intervention (2 months)
Plasma glucose (mg/dL) | Post-intervention (2 months)
  Change in plasma glucose (mg/dL) measured by a blood test from baseline (week 0) to post-intervention (2 months)
Change in total cholesterol (mg/dL) from baseline to post-intervention | Post-intervention (2 months)
  Change in total cholesterol (mg/dL) measured by a blood test from baseline (week 0) to post-intervention (2 months)
Change in total triglycerides (mg/dL) from baseline to post-intervention | Post-intervention (2 months)
  Change in total triglycerides (mg/dL) measured by a blood test from baseline (week 0) to post-intervention (2 months)

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of main findings
Access Criteria: Accepted proposals by the INTERAPNEA-Women team